CLINICAL TRIAL: NCT00002870
Title: A RANDOMIZED, MULTI-CENTRE PHASE III TRIAL TO EVALUATE THE ROLE OF INTENSIFIED THERAPY WITH AUTOLOGOUS TRANSPLANTATION OF HEMATOPOIETIC STEM CELLS IN ADVANCED OR METASTATIC BREAST CANCER RESPONDING TO INDUCTION CHEMOTHERAPY
Brief Title: High Dose Chemotherapy Plus Peripheral Stem Cell Transplantation Compared With Standard Therapy in Treating Women With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PEGASE03; FRE-FNCLCC-PEGASE03; EU-96032
Record Dates: First submitted 1999-11-01; First posted 2004-05-12 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Cyclophosphamide; Epirubicin; Fluorouracil; Thiotepa; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs to kill more tumor cells. It is not yet known if high dose chemotherapy plus peripheral stem cell transplantation is more effective than standard therapy for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of high dose chemotherapy plus peripheral stem cell transplantation with that of standard therapy in treating women who have locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effect on 3-year survival of intensive chemotherapy with cyclophosphamide/thiotepa with peripheral blood stem cell rescue in women with locally recurrent or metastatic breast cancer who respond to induction therapy with epirubicin/fluorouracil/cyclophosphamide. II. Evaluate the effects of this intensive treatment on patient quality of life. III. Evaluate tumor response and progression-free survival after intensification.

OUTLINE: This is a randomized study. Patients are stratified by clinical/therapeutic hormone sensitivity and participating institution. All patients receive induction therapy with epirubicin, fluorouracil, and cyclophosphamide (FEC 100) every 3 weeks for up to 4 courses, with response evaluated after at least 2 courses. Patients with a complete response or at least a 50% partial response are randomized either to no further therapy or to receive intensification chemotherapy. Patients randomized to intensification undergo peripheral blood stem cell (PBSC) harvest with G-CSF mobilization after the third or fourth induction course. Three to 6 weeks after induction, patients receive intensification chemotherapy with cyclophosphamide/thiotepa followed by PBSC. Post-transplant G-CSF is given for hematopoietic support. No concurrent hormonal therapy is permitted during induction; local irradiation of multifocal tumors is allowed provided response is still evaluable. Local therapy (excision of single metastasis, radiotherapy to metastatic site) is permitted after completion of protocol therapy. Treatment of relapsed disease is at the discretion of the investigator. Patients are followed every 3 months for 3 years or until relapse, then every 6 months.

PROJECTED ACCRUAL: A total of 180 patients will be accrued over 3 years in this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven glandular breast cancer Metastatic or locoregionally relapsed disease for which curative surgery and/or radiotherapy is not feasible Histologic/cytologic confirmation of metastasis as feasible Progression required within the month prior to entry, whether or not it occurs on hormonal therapy No clinically detectable cerebral or meningeal involvement Measurable lesion required, including soft tissue site, lymphadenopathy, or visceral site The following are not considered measurable: Bony sites of involvement Ascites Pulmonary lymphangitic carcinomatosis Skin lesions Pathologic CEA or CA 15.3 levels Laboratory changes Pleural effusion Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Under 60 Sex: Women only Menopausal status: Not specified Performance status: WHO 0-2 Life expectancy: Greater than 3 months Hematopoietic: ANC at least 2,000 Platelets at least 100,000 Hepatic: Bilirubin no greater than 2.0 mg/dL (35 micromoles/L) Renal: Creatinine no greater than 1.3 mg/dL (130 micromoles/L) Cardiovascular: No congestive heart failure, even if stable No coronary artery disease No myocardial infarction within 6 months Ventricular ejection fraction (resting) normal by isotopic scan or echocardiogram No evidence of cardiac disease on EKG Other: No active infection No second malignancy except: In situ cervical carcinoma Basal cell skin carcinoma No pregnant women No psychological, familial, social, or geographical contraindication to regular follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior palliative chemotherapy At least 1 year since adjuvant chemotherapy Maximum prior cumulative anthracycline doses as follows: Epirubicin no greater than 450 mg per square meter Doxorubicin no greater than 300 mg per square meter Pirarubicin no greater than 300 mg per square meter Mitoxantrone no greater than 60 mg per square meter Endocrine therapy: Prior hormonal therapy allowed See Disease Characteristics Radiotherapy: At least 6 weeks since radiotherapy to more than one third of hematopoietic regions Surgery: Not specified

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 1994-12; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Biron, MD, Study Chair — Centre Leon Berard
Locations (32):
- France (32):
  - Centre Paul Papin, Angers
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Clinique Saint Vincent, Besançon
  - Institut Bergonie, Bordeaux
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - C.H.U. de Brest, Brest
  - Centre Hospitalier General, Brivé
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Institut Prive de Cancerologie, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Hopital Sainte Blandine, Metz
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Louis, Paris
  - Federation Nationale des Centres de Lutte Contre le Cancer, Paris
  - Hopital Tenon, Paris
  - Hopital Haut Leveque, Pessac
  - Hopital Jean Bernard, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - C.H.U. Saint Etienne Hospital Nord, Saint-Etienne
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Biron P, Durand M, Roche H, Delozier T, Battista C, Fargeot P, Spaeth D, Bachelot T, Poiget E, Monnot F, Tanguy ML, Cure H. Pegase 03: a prospective randomized phase III trial of FEC with or without high-dose thiotepa, cyclophosphamide and autologous stem cell transplantation in first-line treatment of metastatic breast cancer. Bone Marrow Transplant. 2008 Mar;41(6):555-62. doi: 10.1038/sj.bmt.1705935. Epub 2007 Nov 26. PMID 18037940
- [Result] Biron P, Durand M, Roche H, et al.: High dose thiotepa (TTP), cyclophosphamide (CPM) and stem cell transplantation after 4 FEC 100 compared with 4 FEC alone allowed a better disease free survival but the same overall survival in first line chemotherapy for metastatic breast cancer: results of the PEGASE 03 French protocole. [Abstract] Proceedings of the American Society of Clinical Oncology A-167, 2002.